CLINICAL TRIAL: NCT05402774
Title: Abdominal Pain Management and Point-of-care Ultrasound in the Emergency Department: a Randomized, Prospective, Controlled Study
Brief Title: Abdominal Pain Management and Point-of-care Ultrasound in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Necip Gökhan Güner, Emergency Medicine Specialist, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 16214662/050.01.04/152
Record Dates: First submitted 2022-04-18; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Abdominal Pain
Keywords: Abdominal pain; Cost; Emergency department; Length of stay; point-of-care ultrasound
MeSH Terms: conditions — Abdominal Pain; Emergencies

STUDY DESIGN:
Intervention Model Description: a randomized, prospective, controlled study
Who Masked: Care Provider, Outcomes Assessor
Masking Description: At this stage, the patients were divided into two groups: POCUS was applied to patients in the POCUS group after primary clinical evaluation. This procedure was performed in the first hour after the primary clinical evaluations of the patients by evaluating the predetermined parameters in the study form for hepatobiliary, renal, and upper and lower abdominal findings. All processes and results for patients in the control group were followed without any intervention and the results were recorded in the study form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- point-of-care ultrasound group (Other)
  Interventions: Diagnostic Test: point-of-care ultrasound
- Control group (No Intervention)

INTERVENTIONS:
Diagnostic Test: point-of-care ultrasound — point-of-care ultrasound
  Arms: point-of-care ultrasound group

SUMMARY:
Background: Abdominal pain is one of the most common reasons for admission to the emergency department (ED). This study aimed to investigate the effect of point-of-care ultrasound (POCUS) performed during the initial evaluation phase of patients who presented to the ED with abdominal pain on diagnostic processes, length of stay (LOS) in ED, and hospitalization and healthcare costs.

Methodology: This prospective, randomized, controlled, parallel group study was conducted with patients who presented to the Sakarya Education Research Hospital ED with abdominal pain from October 2019 to March 2020. Patients were divided randomly into two groups: control group where standard diagnostic strategies were applied and the POCUS group where POCUS was performed together with standard diagnostic strategies. All data were analyzed using IBM SPSS 21.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* Patients who presented to the ED with abdominal pain
* Nontraumatic patients

Exclusion Criteria:

* permanent mental disability,
* age <18 years,
* abdominal trauma within the last 24 hours,
* pregnancy, morbid obesity, repeated admissions,
* referral from an external center to the ED,
* missing patient information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
to measure the effect of POCUS on the Length of stay in emergency department | 6 months

SECONDARY OUTCOMES:
to measure the effect of POCUS on the average cost of patients, the rate of change in the preliminary diagnosis of the physician, and hospitalization and discharge rate | 1 months after discharge or hospitalisation

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University Training and Research Hospital, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laursen CB, Sloth E, Lassen AT, Christensen Rd, Lambrechtsen J, Madsen PH, Henriksen DP, Davidsen JR, Rasmussen F. Point-of-care ultrasonography in patients admitted with respiratory symptoms: a single-blind, randomised controlled trial. Lancet Respir Med. 2014 Aug;2(8):638-46. doi: 10.1016/S2213-2600(14)70135-3. Epub 2014 Jul 3. PMID 24998674
- [Result] Guner NG, Yurumez Y, Yucel M, Alacam M, Guner ST, Ercan B. Effects of Point-of-care Ultrasonography on the Diagnostic Process of Patients Admitted to the Emergency Department with Chest Pain: A Randomised Controlled Trial. J Coll Physicians Surg Pak. 2020 Dec;30(12):1262-1268. doi: 10.29271/jcpsp.2020.12.1262. PMID 33397050